CLINICAL TRIAL: NCT03845244
Title: Simultaneous Reduction Versus Flow or Fraction of Inspired Oxygen Reduction First in Patients Ready to Wean From High Flow Nasal Cannula Oxygen Therapy: a Randomized Controlled Trial
Brief Title: Weaning Protocol for High Flow Nasal Cannula Oxygen Therapy
Acronym: SLOWH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Sun Kim, Associate professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B-1809-492-006
Record Dates: First submitted 2019-02-11; First posted 2019-02-19 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: High Flow Nasal Cannula; Respiratory Insufficiency
Keywords: high flow nasal cannula; weaning; adult
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Flow reduction first group (Active Comparator): Flow reduction first -> FiO2 reduction -> conventional oxygen therapy
  Interventions: Device: Flow reduction first
- FiO2 reduction first group (Active Comparator): FiO2 reduction first -> flow reduction -> conventional oxygen therapy
  Interventions: Device: FiO2 reduction first
- Simultaneous reduction group (Active Comparator): Simultaneous (Flow and FiO2) reduction -> conventional oxygen therapy
  Interventions: Device: Simultaneous (flow and FiO2) reduction

INTERVENTIONS:
Device: Flow reduction first — -10L/min q 1hr
  Arms: Flow reduction first group
Device: FiO2 reduction first — - 0.1 q 1hr
  Arms: FiO2 reduction first group
Device: Simultaneous (flow and FiO2) reduction — -10L/min and -0.1 q 1hr
  Arms: Simultaneous reduction group

SUMMARY:
High flow nasal cannula oxygen therapy has been widely used in critically ill patients. Despite effectiveness of high flow nasal cannula as a treatment, optimal methods to withdrawal high flow nasal cannula after recovery from preexisting conditions has not been investigated to date. In this study, we will evaluate the efficacy and safety of three different weaning methods in patients with high flow nasal cannula oxygen therapy.

DETAILED DESCRIPTION:
Comparison of three weaning strategies: flow reduction first versus fraction of inspired oxygen (FiO2) first versus simultaneous reduction

ELIGIBILITY:
Inclusion Criteria:

* The patients applying high flow nasal cannula and satisfying the following weaning criteria.

  1. Patient who has recovered from the underlying condition
  2. No signs of respiratory distress like agitation, diaphoresis or anxiety
  3. Arterial pH ≥ 7.35, SpO2 > 90% on FiO2 ≤ 0.5
  4. Respiratory rate ≤ 25/min, Heart rate ≤120/min, Systolic blood pressure ≥ 90mmHg

Exclusion Criteria:

* Severe hypercapnia (pH <7.25)
* Respiratory arrest requiring tracheal intubation
* Cardiac arrest, acute coronary syndrome or life threatening arrhythmias
* Failure of more than two organs
* Recent trauma or burns of the neck and face
* Non- cooperation
* Pregnancy
* Refusal of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Time to weaning success | up to 2 weeks
  The time to successfully remaining off high flow nasal cannula

SECONDARY OUTCOMES:
weaning success or failure rate | up to 2 weeks
  Success or failure rate to wean off high flow nasal cannula
change of arterial partial pressure of oxygen, carbon dioxide, and pH | up to 2 weeks
  changes of arterial blood gas analyses
intolerance rate | up to 2 weeks
  intolerance to high flow nasal cannula
hospital length of stay | during hospital admission, up to 12 weeks
  hospital length of stay
In-hospital mortality | during hospital admission, up to 12 weeks
  all cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Eun Sun Kim, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim MC, Lee YJ, Park JS, Cho YJ, Yoon HI, Lee CT, Lee JH, Kim ES. Simultaneous reduction of flow and fraction of inspired oxygen (FiO2) versus reduction of flow first or FiO2 first in patients ready to be weaned from high-flow nasal cannula oxygen therapy: study protocol for a randomized controlled trial (SLOWH trial). Trials. 2020 Jan 14;21(1):81. doi: 10.1186/s13063-019-4019-7. PMID 31937322